CLINICAL TRIAL: NCT01214538
Title: Assessment of the Natural Antibody Response to Pneumococcal Surface Proteins During Acute Otitis Media in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NasVax Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NX10-07
Record Dates: First submitted 2010-10-03; First posted 2010-10-05 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Acute Otitis Media
Keywords: Vaccine pneumococcal natural history Acute otitis media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group - culture negative: 50 children with pneumococcal culture-negative Acute Otitis Media
- study group- culture positive: 50 children with pneumococcal culture-positive Acute Otitis Media

SUMMARY:
This clinical study is designed to assess prospectively the sero-responses to various proteins in cases of pneumococcal Acute Otitis Media.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Jewish and Bedouin children.
* Patients can be either ambulatory or hospitalized.
* Presenting with acute otitis media.
* Tympanocentesis was performed at least in one ear for a clinical indication.
* Culture of middle ear fluid was obtained.
* Parents agreeing to participate in the study and to submit their children for follow-up, blood test and nasopharyngeal/oropharyngeal (NP/OP) cultures.

Exclusion Criteria:

* Having another infection that is likely to be caused by S. pneumoniae.
* Known immunodeficiency.
* Known previous recent pneumococcal infections (<1 month prior to current visit).

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 100 subjects with acute otitis media infection will be enrolled. The expectation is for ≥50 children with pneumococcal culture-positive MEF (Middle Ear Fluid) and ≥50 children with culture-negative MEF to be enrolled
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-03 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Serological studies of pneumococcal proteins and their development over time following otitis media infections | 3 months per individual
  The serological studies will study the natural immune response to protective pneumococcal vaccine antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Dagan, Prof. MD., Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Ben-Gurion University of the Negev, Beersheba, Israel